CLINICAL TRIAL: NCT01456819
Title: Phase II Efficacy Study of Intramuscular Autologous Bone Marrow Mononuclear Cells Plus Mesenchymal Stem Cell Implantation Versus Autologous Bone Marrow Mononuclear Cells Implantation Only in Patients With Chronic Critical Limb Ischemia
Brief Title: Intramuscular Mononuclear Cells and Mesenchymal Stem Cells Transplantation to Treat Chronic Critical Limb Ischemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Cytopeutics Sdn. Bhd. (Industry)
Responsible Party: Principal Investigator, Dr Hanafiah Harunarashid, Senior Consultant Vascular Surgeon, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FF-113-2011; NMRR-11-904-9763 (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2011-10-04; First posted 2011-10-21 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Critical Limb Ischemia
Keywords: autologous; bone marrow; critical limb ischemia; efficacy; mesenchymal stem cells; mononuclear cells
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mononuclear and mesenchymal stem cells (Experimental): Autologous bone marrow-derived mononuclear cells and mesenchymal stem cells
  Interventions: Biological: Mononuclear and mesenchymal stem cells
- Mononuclear cells only (Active Comparator): Autologous bone marrow-derived mononuclear cells
  Interventions: Biological: Mononuclear cells

INTERVENTIONS:
Biological: Mononuclear and mesenchymal stem cells — Intramuscular administration into the ischemic limb
  Other Names: BM-MNC and BM-MSC
  Arms: Mononuclear and mesenchymal stem cells
Biological: Mononuclear cells — Intramuscular administration into the ischemic limb
  Other Names: BM-MNC
  Arms: Mononuclear cells only

SUMMARY:
This is a randomized and single blinded study aimed to compare the efficacy between intramuscular autologous bone marrow mononuclear cells plus mesenchymal stem cell implantation and intramuscular autologous bone marrow mononuclear cells implantation only in patients with chronic critical limb ischemia. Patients will be randomized into two groups of equal number; patients in one group will be implanted with mononuclear cells and mesenchymal stem cells, and the other implanted with mononuclear cells only in the area of affected limb.

DETAILED DESCRIPTION:
When the long blood vessels supplying blood to the arms and legs become blocked (ischemic), patient will experience painful sensations in their calves when they walked which slowly become excruciating painful at rest. When the condition worsens, the patients will not be able to feel any pain from their legs and they will not know if there are any small ulcers or cuts on their legs. As a result, a small ulcer which goes unnoticed becomes bigger and can sometimes become infected. In the worst situations, infection might lead towards gangrene and septicaemia. Severe rest pain and/or ulcerations of ischemic limbs are defined as the state of chronic critical limb ischemia and at this point, amputation of the affected limb is suggested.

Conventional treatments include angioplasty/bypass operation to remove blood vessel blockage to restore blood supply, the use of prescribed medicines to aid in ulcer recovery and clear infection and debridement of damaged/infected tissue. Some procedures have to be performed multiple times. Amputation is inevitable in many cases because some blood capillaries cannot be corrected and restenosis of vessels is very common. Cell therapy with mononuclear cells and mesenchymal stem cells from bone marrow is promising because these stem cells are capable of stimulating and regenerating capillaries and blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of critical limb ischemia leading to ischemic ulcers in which amputation is indicated
* Not suitable for, or remain symptomatic despite angioplasty, bypass operation or collateralization

Exclusion Criteria:

* Contraindication to epidural anesthesia and bone marrow aspiration
* Contraindication to contrast angiography
* Evidence of neoplasia and bone marrow diseases
* Any acute or chronic communicable diseases including Hepatitis B, Hepatitis C and HIV
* Patients with a limited life expectancy (< 1 year)
* Patients with myocardial infarction or stroke within 6 months
* Patients with coronary intervention within 6 months
* Renal impairment indicated by serum creatinine greater than two times upper limit of the normal range
* Liver impairment indicated by serum aspartate transaminase and alanine transaminase greater than two times upper limit of normal
* Any other co-morbidity which the physician deems as a contraindication to stem cell transplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in angiogenesis | 1 month, 3 months, 6 months, 9 months, 12 months
  Measurement of angiogenesis by presence of peripheral pulses, capillary refill and transcutaneous oxygen saturation (TCOS).

SECONDARY OUTCOMES:
Change in ulcer size | 1 month, 3 months, 6 months, 9 months, 12 months
  Measurement of ulcer size by clinical assessment and grid maps.
Visual Analog Score | 1 month, 3 months, 6 months, 9 months, 12 months
Exercise Treadmill Test | 1 month, 3 months, 6 months, 9 months, 12 months
Improvement in vascularity and blood supply | 1 month, 3 months, 6 months, 9 months and 12 months
  Measured by digital subtraction angiography (DSA) and ankle brachial systemic pressure index (ABI).

CONTACTS AND LOCATIONS:
Overall Officials: Hanafiah Harunarashid, MD, Principal Investigator — UKM Medical Centre
Locations (1):
- UKM Medical Centre, Kuala Lumpur, Malaysia